CLINICAL TRIAL: NCT01700322
Title: Effects of Clopidogrel vs Prasugel vs Ticagrelor on Endothelial Function, Inflammatory and Oxidative Stress Parameters and Platelet Function in Patients Undergoing Coronary Artery Stenting. A Randomised, Prospective Study.
Brief Title: Endothelium, Stenting, and Antiplatelet Therapy (EST) - Clopidogrel, Prasugrel, Ticagrelor Study
Acronym: EST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Tommaso Gori, Professor, Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: CTH-C1
Record Dates: First submitted 2012-09-04; First posted 2012-10-04 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; coronary stenting; platelet aggregation
MeSH Terms: conditions — Coronary Artery Disease | interventions — Ticagrelor; Clopidogrel; Prasugrel Hydrochloride

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ticagrelor (Active Comparator): Ticagrelor 180mg oral loading dose and 90mg b.i.d for 30 days following coronary artery stenting
  Interventions: Procedure: Coronary stenting; Drug: Ticagrelor
- Clopidogrel (Active Comparator): Clopidogrel 600mg loading dose + 75 mg once a day for 30 days following coronary artery stenting.
  Interventions: Procedure: Coronary stenting; Drug: Clopidogrel
- Prasugrel (Active Comparator): Prasugrel 60mg oral loading dose followed by 10mg once a day for 30 days following coronary artery stenting
  Interventions: Procedure: Coronary stenting; Drug: Prasugrel

INTERVENTIONS:
Procedure: Coronary stenting — All patients will receive a drug eluting stent as clinically indicated.
Drug: Ticagrelor — Ticagrelor 180mg oral loading dose and 90mg b.i.d for 30 days following coronary artery stenting
  Arms: Ticagrelor
Drug: Clopidogrel — Clopidogrel 600mg loading dose + 75 mg once a day for 30 days following coronary artery stenting.
  Arms: Clopidogrel
Drug: Prasugrel — Prasugrel 60mg oral loading dose followed by 10mg once a day for 30 days following coronary artery stenting
  Arms: Prasugrel

SUMMARY:
Endothelial dysfunction is an important predictor - and a determinant - of adverse clinical outcome. Endothelial function is impaired by coronary artery stenting, a stud from our group has shown that it can be improved by platelet inhibition using clopidogrel. However, clopidogrel unresponsiveness is a known problem, and it has been show that the endothelial effects of clopidogrel tend to wane upon prolonged treatment. Whether a more effective anti-platelet therapy is able to prevent/improve not only thrombotic events but also endothelial dysfunction, with potential positive impact on clinical outcome in patients undergoing coronary artery stenting, is an important hypothesis that needs to be further investigated. To date, evidence regarding "ancillary" (non-platelet-dependent) effects of antiaggregant drugs is very limited. For instance, while their antiplatelet effects, and their beneficial effects in patients with acute coronary syndromes, have been clearly demonstrated in multicentric trials, it remains to be shown whether these drugs also protect endothelial function. Interestingly, some authors suggest that the mortality benefit observed in the PLATO study is at least in part independent of direct antiplatelet effects. No study, to date, has tested the effects of prasugrel and/or ticagrelor on endothelial function. With the present trial, the investigators plan to test the effect of clopidogrel, prasugrel and ticagrelor on endothelial function before and up to 4 weeks after coronary artery stenting. This study will provide important pathophysiologic insight on the relationship between platelet aggregation and endothelial function, two parameters that have been shown to influence patients' prognosis.

ELIGIBILITY:
Inclusion Criteria:

* - 18-75 years old consecutive patients undergoing coronary angiography and stenting at the University Medical Centre Mainz
* A coronary lesion (and patient) amenable to treatment with drug eluting stent
* Ability of subject to understand character and individual consequences of clinical trial
* Signed and dated informed consent of the subject must be available before start of any specific trial procedures.
* Negative pregnancy test of women with childbearing potential

Exclusion Criteria:

* Subjects presenting 1 or more of the following criteria will not be enrolled in the trial:
* Patients with elevated (> 5 times upper normal limit) C-reactive protein level prior to stenting
* Patients in whom therapy with long-acting nitrates cannot be suspended prior to endothelial function measurements
* An acute coronary syndrome treated with coronary stenting within the last 4 weeks
* Patients with known inflammatory/infective diseases
* Patients with severe extracardiac diseases limiting life expectancy
* Known heart failure (LV-EF ≤ 40% AND NYHA III-IV)
* PCI or coronary By-Pass surgery within the last 4 weeks, pre-existing ongoing treatment with any of the study treatments.
* History of cerebrovascular events (stroke)
* Known renal dysfunction (serum creatinine ≥ 1.8mg/dl in women, ≥ 2.0mg/dl in men)
* Serum potassium > 5.5mmol/l
* Known hepatic impairment (AST, ALT > 3 times upper limit of normal)
* Changes in the ß-blocker, statin or ACE or angiotensin-receptor blocker inhibitor treatment within the past 2 weeks
* Pregnancy and lactation, inadequate contraception
* Body weight < 60kg
* Active bleeding
* Therapy with CYP3A4 inhibitors (ketoconazole, protease inhibitors, macrolide antibiotics)
* Therapy with anticoagulants: phenprocoumone, warfarin, dabigatran, rivaroxaban
* History of hypersensitivity to any of the investigational medicinal products or to any drug with similar chemical structure or to any excipient present in the pharmaceutical form of the investigational medicinal product.
* Ongoing participation in other clinical trials or within the last 3 months, or ongoing therapy with one of the study medications.
* Medical or psychological condition that would not permit completion of the trial or signing of informed consent.
* Patients with acute ST-elevation myocardial infarction

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2012-08; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in FMD | baseline and 1 month
  The primary endpoint is the change in flow-mediated dilation (FMD) (comparison before treatment versus after treatment and stenting) in the three study groups. The mean FMD across the three measurements (1 day, 1 week, 1 month) performed after coronary artery stenting will be compared to the FMD value before drug administration and stenting.

SECONDARY OUTCOMES:
FMD 2 hours after loading dose | baseline and 2 hours after loading dose
  Change in FMD 2 hours after the administration of the study drug
L-FMC at 2 hours after the loading dose | baseline and 2 hours
  change in L-FMC at two hours after the loading dose
L-FMC 1 month after loading dose | baseline and 1 day after stenting
  change in flow-mediated constriction (L-FMC) (comparison before treatment versus after treatment and stenting) in the three study groups. The mean L-FMC across the three measurements (1 day, 1 week, 1 month) performed after coronary artery stenting will be compared to the value before drug administration and stenting
Safety and tolerability | from baseline to 1 month after enrollment
  Number of patients with adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Munzel, MD Prof., Study Chair — University Medical Center Mainz
Locations (1):
- 2 Medical Clinic, Mainz, Germany

REFERENCES:
- [Derived] Schnorbus B, Jurk K, Lackner KJ, Welk C, Munzel T, Gori T. Effects of Clopidogrel, Prasugrel and Ticagrelor on Microvascular Function and Platelet Reactivity in Patients With Acute Coronary Syndrome Undergoing Coronary Artery Stenting. A Randomized, Blinded, Parallel Group Trial. Front Cardiovasc Med. 2021 Dec 13;8:780605. doi: 10.3389/fcvm.2021.780605. eCollection 2021. PMID 34966798
- [Derived] Schnorbus B, Daiber A, Jurk K, Warnke S, Konig J, Krahn U, Lackner K, Munzel T, Gori T. Effects of clopidogrel, prasugrel and ticagrelor on endothelial function, inflammatory and oxidative stress parameters and platelet function in patients undergoing coronary artery stenting for an acute coronary syndrome. A randomised, prospective, controlled study. BMJ Open. 2014 May 6;4(5):e005268. doi: 10.1136/bmjopen-2014-005268. PMID 24801283